CLINICAL TRIAL: NCT06293638
Title: Functional Brain Network Changes in Patients Undergoing Deep Brain Stimulation for Essential Tremor
Acronym: TRaNCE
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, James Liao, Principal Investigator, The Cleveland Clinic
Other Study IDs: 23-1125
Record Dates: First submitted 2024-01-30; First posted 2024-03-05 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor
Keywords: essential tremor; deep brain stimulation; DBS; ET; tremor; hand tremors
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Ethanol; Alprazolam; Cryotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Essential Tremor with DBS: 1. 30-80 years of age
  2. Diagnosis of ET
  3. Previously implanted with a DBS system for disease management per standard of care
  Interventions: Drug: Alcohol; Drug: Alprazolam; Device: Cold Therapy; Procedure: Peripheral Nerve Stimulation
- Essential Tremor without DBS: 1. 30-80 years of age
  2. Diagnosis of ET
  3. Has not been previously implanted with a DBS system for disease management per standard of care
  Interventions: Drug: Alcohol; Drug: Alprazolam; Device: Cold Therapy; Procedure: Peripheral Nerve Stimulation
- No Known Neurological Disease or Disorder: 1. 30-80 years of age
  2. No known neurological disease or disorder
  Interventions: Drug: Alcohol; Drug: Alprazolam; Device: Cold Therapy; Procedure: Peripheral Nerve Stimulation

INTERVENTIONS:
Drug: Alcohol — Alcohol consumption is shown to reduce tremor in individuals with essential tremor. The alcoholic beverage will be dispensed by the a clinician study investigator, and the participant will be administered the alcoholic beverage until their tremor is decreased, as determined by the clinician. Individual sensitivity to the tremor-mitigating effects of alcohol varies, but it is anticipated that only light (1-2 40% ABV drinks, containing 1-2 units of absolute alcohol [10 mL. or 8 g of pure ethanol]) consumption will be necessary. Participants will then repeat motor task and data collection while the alcohol is effective at controlling tremor, beginning approximately 15-20 minutes after consumption.
  Other Names: Vodka
Drug: Alprazolam — Alprazolam is shown to reduce tremor in individuals with essential tremor. The primary investigator will select the appropriate dose for the patient (0.5mg for patients with a body weight of up to 75kg, and 0.75mg for participants with a body weight of 75kg and higher). Participants will swallow the drug with a glass of water in the presence of the research team. If participants have not reached a sufficient level of tremor improvement, a subsequent dose of up to a total of 1.0mg of alprazolam per participant will be requested. Participants will then repeat motor task and data collection.
  Other Names: Xanax
Device: Cold Therapy — One or both of the participant's upper limbs will be wrapped with pre-chilled ice packs or a cold water circulating device such as a cryomanchet (e.g., the Breg PolarCare Glacier), and the skin temperature monitored until it lowers to 15-25°C. Participants will then repeat motor task and data collection while the limb is cool.
  Other Names: BREG Polar Care Glacier Cold Therapy System
Procedure: Peripheral Nerve Stimulation — Electrical stimulation will be applied using techniques similar to those applied during standard somatosensory evoked potential testing. Specifically, adhesive surface electrodes will be placed above the median and radial nerves at the wrist. Stimulation paradigms will be tailored to each participant based on the frequency characteristics of their tremor. Participants will receive between 20-60 minutes of stimulation, then will repeat motor task and data collection. Transcutaneous peripheral nerve stimulation may help mitigate tremor, with effects lasting beyond cessation of stimulation1-3.

SUMMARY:
The purpose of this study is to collect electrophysiological data related to functional brain network changes in patients undergoing deep brain stimulation for the treatment of essential tremor. Participants will either 1) have electroencephalography (EEG) scalp electrodes placed, or 2) remain seated with their head inside of a magnetoencephalography (MEG) recording system, as resting-state and task-related data are acquired. Spontaneous electrophysiological activity will be recorded in both the eyes open and eyes closed conditions with the participant seated comfortably. These recordings will be repeated in the DBS OFF and DBS ON states, with the ON state involving specific settings identified as optimal, sub-optimal, or ineffective at achieving tremor control. They will also be repeated following the optional administration non-DBS tremor mitigation techniques, which may include one or more of the following: 1) cooling the limb, 2) oral administration of alprazolam, 3) oral consumption of ethanol (alcohol), or 4) peripheral nerve stimulation.

DETAILED DESCRIPTION:
Electrophysiological data from participants will be collected during electroencephalography (EEG) or magnetoencephalography (MEG) procedures. The EEG or MEG experiments will also include recordings from the DBS system that may be synchronized to externally recorded signals (e.g., MEG, EEG, EMG, accelerometry) via gentle tap-induced motion artifacts, and/or by applying a small, barely perceptible electrical current at the skin over the DBS system with use of a transcutaneous electrical nerve stimulation (TENS) unit.

It is hypothesized that the chronic, electrical stimulation of the target region has both local and circuit-wide effects, the net effect of which is to disrupt the pathophysiological neural activity present across both cortical and subcortical brain regions that and thought to underlie disease manifestation (i.e., tremor). By systemically characterizing the pathways involved in propagating tremor-related activity as well as mediating treatment-related benefits, the investigators hope to identify potential new therapeutic targets or treatment paradigms to further optimize tremor control in this population.

ELIGIBILITY:
Inclusion Criteria:

* Between 30 and 80 years of age;
* Ability to provide informed consent;
* Clinical diagnosis of ET by a movement disorders neurologist with a disease duration of at least 3 years and being treated with a DBS; OR
* Clinical diagnosis of ET by a movement disorders neurologist with a disease duration of at least 3 years and not being treated with a DBS; OR
* No known neurological disease or disorder.

Exclusion Criteria:

* The individual has a condition that, in the opinion of the investigator, would significantly increase the risk for interference with study compliance, safety, or outcome;
* Presence of active psychiatric symptoms meeting Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for Axis-I disorder on formal psychiatric evaluation other than depression or anxiety;
* History of cognitive impairment meeting Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for dementia on formal neuropsychological evaluation, as documented in chart;
* Lack of English-language fluency which would interfere with the ability to understand the study consenting process and potential study risks;
* Hearing or visual impairment precluding testing;
* Motor impairment impacting test responses (i.e., orthopedic injury or disease);
* Anyone currently taking medications with Antabuse-like effects (e.g. Flagyl, Bactrim, Tindamax) will be excluded from any alcohol administration.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the known patient population from a large research medical center located in a medium-to-large American city.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CTCM Coherence | up to 8 hours in-lab during experiment
  Coherence, a unitless measure of correlation between signals, calculated across the cerebellothalmocorticomuscular (CTCM) circuit, will be computed from neurophysiological recordings including electroencephalography (EEG), electromyography (EMG), magnetoencephalography (MEG), and/or local field potential (LFP), using data collected at rest, during tremor-eliciting tasks, with DBS OFF, with DBS ON (when available), and when using non-DBS tremor interventions (limb cooling and/or peripheral nerve stimulation and/or alprazolam or alcohol).
Power of oscillatory activity across the CTCM network in response to tremor interventions | up to 8 hours in-lab during experiment
  Power of tremor-related oscillatory activity, in the form of mean power in the 4-12Hz frequency band with units in mV^2, will be computed from neurophysiological recordings including electroencephalography (EEG), electromyography (EMG), magnetoencephalography (MEG), and/or local field potential (LFP), using data collected at rest, during tremor-eliciting tasks, with DBS OFF, with DBS ON (when available), and when using non-DBS tremor interventions (limb cooling and/or peripheral nerve stimulation and/or alprazolam or alcohol).

SECONDARY OUTCOMES:
Essential tremor severity: Limb acceleration | up to 8 hours in-lab during experiment
  Accelerometers placed on the limb will measure tremor energy in the 4-12Hz band, in units of mG^2/Hz. Data is collected at rest, during tremor-eliciting tasks, with DBS OFF, with DBS ON (when available), and when using non-DBS tremor interventions (limb cooling and/or peripheral nerve stimulation and/or alprazolam or alcohol).
Essential tremor severity: Tremor Research Group Essential Tremor Rating Scale (TETRAS) | up to 8 hours in-lab during experiment
  Numerical clinical tremor assessment scale correlated with severity of tremor. Data is collected with DBS OFF, with DBS ON (when available), and when using non-DBS tremor interventions (limb cooling and/or peripheral nerve stimulation and/or alprazolam or alcohol). Items are scored 0-4 with "0" being normal and "4" being severely abnormal.
Essential tremor severity: Grip force | up to 8 hours in-lab during experiment
  A hand-held force sensor will measure grip force (Newtons). Data is collected at rest, during tremor-eliciting tasks, with DBS OFF, with DBS ON (when available), and when using non-DBS tremor interventions (limb cooling and/or peripheral nerve stimulation and/or alprazolam or alcohol).

CONTACTS AND LOCATIONS:
Overall Officials: James Liao, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No